CLINICAL TRIAL: NCT00307073
Title: Adapta Clinical Study to Evaluate the Overall System Safety and Clinical Performance of the Adapta Pacing System
Brief Title: Adapta Pacing System Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201
Record Dates: First submitted 2006-03-17; First posted 2006-03-27 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Pacemaker; Bradycardia
Keywords: Pacemaker; Managed Ventricular Pacing; Ventricular Pacing
MeSH Terms: conditions — Bradycardia

INTERVENTIONS:
Device: Implantable Pulse Generator

SUMMARY:
Pacemakers are implantable devices that pace (electrically stimulate) the heart. Some pacemakers have special programs to treat irregular atrial rhythms(top chambers of the heart beat too fast or too slow). Advances in pacemaker technology in recent years include features that automatically adapt to patient conditions without intervention from the clinician. Adapta (Model #ADDR01) is a new pacemaker that is designed to provide further automaticity advances by including the managed ventricular pacing (MVP) feature designed to promote intrinsic conduction (natural flow of electricity in the heart) by reducing unnecessary ventricular (lower chamber of the heart) pacing (electrical impulses). Adapta also contains a feature called TherapyGuide that is designed to allow the user to select certain conditions for each subject and receive a list of suggested pacemaker parameter value changes based on those conditions. The purpose of this study is to evaluate the overall system safety and clinical performance of the Adapta pacing system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a Class I or II indication for implantation of a dual chamber pacemaker according to ACC/AHA/NASPE guidelines
* Subjects who have signed a Medical Ethics Committee (MEC) approved Informed Consent Form

Exclusion Criteria:

* Subjects with a mechanical tricuspid valve
* Subjects with a life expectancy less than two years
* Subjects with a Class III indication for permanent pacing
* Subjects with lead integrity problems, unless leads are being replaced

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2005-05; Study Completion 2005-11

PRIMARY OUTCOMES:
Freedom from adverse device effects

SECONDARY OUTCOMES:
To assess right ventricular (lower right chamber of the heart) pacing
To summarize all adverse events reported in the study
To describe Adapta system performance as observed during Holter recording, save-to disk-files and technical observations
To evaluate the user acceptance of TherapyGuide via questionnaire data

CONTACTS AND LOCATIONS:
Overall Officials: Adapta Study Team, Study Chair — Medtronic
Locations (7):
- Graz, Austria
- Prague, Czechia
- Germany (2):
  - Bad Nauheim
  - Hamburg
- Heerlen, Netherlands
- Belgrade, Serbia and Montenegro
- Lund, Sweden